CLINICAL TRIAL: NCT04098588
Title: Behavioral Economics Intervention to Increase Treatment Seeking in the National Guard
Acronym: BEAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern Mississippi (Other)
Collaborators: Military Suicide Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-16-2-0003
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Treatment Refusal
MeSH Terms: conditions — Treatment Refusal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEAST (Experimental): There are 3 parts to BEAST. Part 1 involves the Behavioral Nudge technique using previously collected injunctive and descriptive norms from a National Guard sample. Soldiers will be given a customized feedback form that shows norms relevant to the target behavior they selected. The soldier will be given a chance to ask any follow-up questions. Part 2 of the intervention focuses on the principle of targeting others, considering how a change would impact those closest to them. Part 3 will utilize the Reciprocal Concessions procedure combined with the Reducing Barriers technique.
  Interventions: Behavioral: BEAST
- Descriptive Feedback (Active Comparator): This condition will involve a presentation of descriptive data based on the soldiers' tests scores and an opportunity to ask any follow-up questions. This process is a component of some behavioral change interventions (e.g., motivational interviewing); therefore this should be a more useful control condition (mirroring parts 1 and 2 of the active condition) versus a more passive or waitlist control condition. Participants in the control condition will also be given standard referral information to the USM Psychology Clinic (mirroring part 3 of the active condition).
  Interventions: Behavioral: Descriptive Feedback

INTERVENTIONS:
Behavioral: BEAST — See Arm Description
  Arms: BEAST
Behavioral: Descriptive Feedback — See Arm Description
  Arms: Descriptive Feedback

SUMMARY:
The study is a randomized controlled trial of a single-session behavioral economics (research combining the areas of economics, social psychology, and cognitive psychology) intervention (i.e., BEAST) is a"warrior-culture" consistent (i.e., focusing on positive soldier traits, solving practical problems), highly scalable, and extremely brief (10-minute) intervention to encourage treatment seeking among MS National Guard problems for various life stressors. Participants will be 112 National Guard members. It is hypothesized that BEAST will lead to more self-reported motivation to seek treatment and more actual treatment seeking behavior.

ELIGIBILITY:
Inclusion Criteria:

* National Guard active
* > 17 ACSS-FAD

Exclusion Criteria:

* those determined by military or study personnel to be actively psychotic, manic, or who are imminently suicidal and in need of emergency services.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2023-03-29 (Estimated); Study Completion 2023-03-29 (Estimated)

PRIMARY OUTCOMES:
Psychosocial Treatments Interview-Revised | 1 month post intervention
  Measure changes in treatment seeking behavior
University of Rhode Island Change Assessment | 1 month post intervention
  Measure motivation to change the target behavior

SECONDARY OUTCOMES:
Psychosocial Treatments Interview-Revised | 3 month post intervention
  Measure changes in treatment seeking behavior
University of Rhode Island Change Assessment | 3 month post intervention
  Measure motivation to change the target behavior

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Undecided
After the study is completed will discuss with Department of Defense /Military Suicide Research Consortium on ability to share IPD.